CLINICAL TRIAL: NCT01152450
Title: A Phase II, Randomised, Double- Blind, Placebo Controlled, Cross-over Efficacy and Safety Comparison of Tiotropium 5 µg Administered Once Daily (in the Evening) and Tiotropium 2.5 µg Administered Twice Daily Delivered by the Respimat® Inhaler for Four Weeks Versus Placebo in Patients With Moderate Persistent Asthma
Brief Title: A Randomised, Double- Blind, Placebo Controlled, Cross-over Efficacy and Safety Comparison of Tiotropium 5 µg Once Daily and Tiotropium 2.5 µg Twice Daily for Four Weeks in Patients With Moderate Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.420; 2009-018006-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (3):
- Tiotropium daily dose q.d. (Experimental): two actuations delivered via Respimat® inhaler
  Interventions: Drug: Tiotropium 5 µg q.d.
- Tiotropium half daily dose b.i.d. (Experimental): two actuations delivered via Respimat® inhaler
  Interventions: Drug: Tiotropium 2.5 µg b.i.d
- Placebo (Placebo Comparator): N/A (two actuations of placebo) delivered via Respimat® inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium 2.5 µg b.i.d — 2.5 µg (two actuations of 1.25 µg) delivered via Respimat® inhaler
  Arms: Tiotropium half daily dose b.i.d.
Drug: Placebo — N/A (two actuations of placebo) delivered via Respimat® inhaler
  Arms: Placebo
Drug: Tiotropium 5 µg q.d. — 5 µg (two actuations of 2.5 µg) delivered via Respimat® inhaler
  Arms: Tiotropium daily dose q.d.

SUMMARY:
Rationale for the current trial is to demonstrate 24 hour bronchodilator efficacy and safety of tiotropium 5 µg administered once daily (in the evening) which is regarded beneficial for the compliance and convenience of the patient in comparison to placebo. Further the rationale is to evaluate efficacy and safety of tiotropium 2.5 µg administered twice daily delivered by the Respimat® inhaler in comparison to placebo and tiotropium 5 µg administered once daily (in the evening) delivered by the Respimat® inhaler in patients with moderate persistent asthma.

Rationale for the pharmacokinetic subinvestigation is to evaluate the 24 hours exposure to tiotropium in patients with moderate persistent asthma when administered 5 µg tiotropium once daily (in the evening) or 2.5 µg tiotropium twice daily.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign and date an Informed Consent Form consistent with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice ( ICH-GCP) guidelines and local legislation prior to participation in the trial (i.e. prior to any trial procedures, including any pre-trial washout of medications and medication restrictions for pulmonary function test at Visit 1).
2. Male or female patients aged at least 18 years but not more than 75 years.
3. All patients must have at least a 3 months history of asthma at the time of enrolment into the trial. The diagnosis of asthma has to be confirmed at Visit 1 with a bronchodilator reversibility resulting in a Forced Expiratory Volume in 1 Second (FEV1) increase of equal above 12% and equal above 200mL.
4. The initial diagnosis of asthma must have been made before the patient's age of 40.
5. All patients must have a diagnosis of moderate persistent asthma and must be symptomatic despite their current maintenance treatment with medium doses of inhaled corticosteroids.
6. All patients must have been on maintenance treatment with a medium, stable dose of inhaled corticosteroids (alone or in a fixed combination with a Long Acting Betaadrenergic (LABA) or Short Acting Betaadrenergic (SABA)) for at least 4 weeks prior to Visit 1.
7. All patients must be symptomatic at Visit 1 (screening) and Visit 2 as defined by an Asthma Control Questionnaire (ACQ) Score
8. All patients must have a pre-bronchodilator FEV1 above equal 60% predicted and below equal 90% of predicted normal at Visit 1. Predicted normal values will be calculated according to the European Coal and Steel Community Guidelines (ECSC).
9. All patients must have an increase in FEV1 of equal above 12% and equal above 200 mL 15 minutes after 400 µg salbutamol at Visit 1.
10. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator) as compared to Visit 2 (pre-dose) must be within ± 30% .
11. Patients must be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment and who have a smoking history of less than 10 pack years.
12. Patients must be able to use the Respimat® inhaler correctly.
13. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of the e-Diary/peak flow meter.
14. Patients taking a chronic pulmonary medication allowed by the study protocol must be willing to continue this therapy for the entire duration of the study (exception: times of acute disease deterioration).

Exclusion criteria:

1. Patients with a significant disease other than asthma.A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
2. Patients with a clinically relevant abnormal screening hematology or blood chemistry if the abnormality defines a significant disease as defined in exclusion criterion no. 1.
3. Patients with a recent history (i.e. six months or less) of myocardial infarction.
4. Patients who have been hospitalised for cardiac failure during the past year.
5. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
6. Patients with lung diseases other than asthma (e.g. Chronic Obstructive Lung Disease (COPD)).
7. Patients with known active tuberculosis.
8. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed.
9. Patients who have undergone thoracotomy with pulmonary resection.
10. Patients with significant alcohol or drug abuse within the past two years.
11. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to V 1.
12. Patients with known hypersensitivity to anticholinergic drugs, Benzalconiumchloride (BAC), Ethylenediaminetetraacetate (EDTA) or any other components of the study medication delivery systems.
13. Pregnant or nursing women.
14. Women of childbearing potential not using a highly effective method of birth control.
15. Patients who have been treated with beta-blocker medication within four weeks prior to Visit 1 or during the screening period. Topical cardio-selective beta-blocker eye medications for non-arrow angle glaucoma are allowed.
16. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva®) within four weeks prior to Visit 1 or during the screening period.
17. Patients who have been treated with oral beta-adrenergics within four weeks prior to Visit 1 or during the screening period.
18. Patients who have been treated with oral corticosteroids within four weeks prior to Visit 1 or during the screening period.
19. Patients who have been treated with anti-IgE antibodies, e.g. omalizumab (Xolair®), within 6 months prior to Visit 1 or during the screening period.20. Patients who have been treated with cromolyn sodium or nedocromil sodium within two weeks prior to Visit 1 or during the screening period.

21. Patients who have been treated with methylxanthines within two weeks prior to Visit 1 or during the screening period.

22. Patients who have taken an investigational drug within four weeks prior to Visit 1.

23. Patients who have been treated with other non-approved and according to international guidelines not recommended "experimental" drugs for routine asthma therapy (e.g. TNFalpha blockers, methotrexate, cyclosporin) within four weeks prior to Visit 1 or during the screening period.

24. Patients with any asthma exacerbation or any respiratory tract infection in the four weeks prior to Visit 1 or during the screening period. Visit 1 and/or Visit 2 should be postponed in case of an asthma exacerbation or respiratory tract infection.

25. Patients who have previously been randomised in this trial or are currently participating in another trial.

26.Patients who have been treated with depot corticosteroids within six months prior to Visit 1 or during the screening period.

27.Patients who have been treated with leukotriene modifiers within two weeks prior to Visit 1 or during the screening period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- Austria (4):
  - 205.420.43002 Boehringer Ingelheim Investigational Site, Linz
  - 205.420.43004 Boehringer Ingelheim Investigational Site, Schlüsslberg
  - 205.420.43003 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
  - 205.420.43001 Boehringer Ingelheim Investigational Site, Wels
- Czechia (2):
  - 205.420.42002 Boehringer Ingelheim Investigational Site, Brno
  - 205.420.42001 Boehringer Ingelheim Investigational Site, Kyjov
- Estonia (2):
  - 205.420.37201 Boehringer Ingelheim Investigational Site, Kohtla-Järve
  - 205.420.37202 Boehringer Ingelheim Investigational Site, Tallinn
- Germany (4):
  - 205.420.49002 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 205.420.49004 Boehringer Ingelheim Investigational Site, Hanover
  - 205.420.49001 Boehringer Ingelheim Investigational Site, Mannheim
  - 205.420.49003 Boehringer Ingelheim Investigational Site, Schwerin
- Latvia (3):
  - 205.420.37102 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.420.37101 Boehringer Ingelheim Investigational Site, Riga
  - 205.420.37103 Boehringer Ingelheim Investigational Site, Riga

REFERENCES:
- [Derived] Timmer W, Moroni-Zentgraf P, Cornelissen P, Unseld A, Pizzichini E, Buhl R. Once-daily tiotropium Respimat((R)) 5 mug is an efficacious 24-h bronchodilator in adults with symptomatic asthma. Respir Med. 2015 Mar;109(3):329-38. doi: 10.1016/j.rmed.2014.12.005. Epub 2014 Dec 27. PMID 25661281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 94 patients entered the study and was treated whilst 89 patients completed the trial.
Pre-assignment Details: Randomised, double-blind, placebo controlled, cross-over design without washout phase between the three periods. Patients were randomized equally to one of the six sequences (ABC, ACB, BAC, BCA, CAB, CBA).
Groups:
- Tio R2.5 Twice Daily (Bid) /Tio R5 Once Daily (qd) /Placebo: Patients treated with Tiotropium 2.5 mcg in period 1 (morning and evening), with a matching placebo in the morning and Tiotropium 5 mcg in the evening in period 2 and with a matching Placebo in period 3 (morning and evening). All products were delivered by the Respimat inhaler, on top on maintenance therapy with inhaled corticosteroid (iCS). No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Tio R2.5 Bid/Placebo/Tio R5 qd: Patients treated with Tiotropium 2.5 mcg in period 1 (morning and evening), with a matching Placebo in period 2 (morning and evening) and with a matching placebo in the morning and Tiotropium 5 mcg in the evening in period 3. All products were delivered by the Respimat inhaler, on top on maintenance therapy with iCS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Tio R5 qd/Tio R2.5 Bid/Placebo: Patients treated with a matching placebo in the morning and Tiotropium 5 mcg in the evening in period 1, with Tiotropium 2.5 mcg in period 2 (morning and evening) and with matching Placebo in period 3 (morning and evening) . All products were delivered by the Respimat inhaler, on top on maintenance therapy with iCS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Tio R5 qd/Placebo/Tio R2.5 Bid: Patients treated with a matching placebo in the morning and Tiotropium 5 mcg in the evening in period 1, with matching Placebo in period 2 (morning and evening) and with Tiotropium 2.5 mcg in period 3 (morning and evening) . All products were delivered by the Respimat inhaler, on top on maintenance therapy with iCS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Placebo/Tio R2.5 Bid/Tio R5 qd: Patients treated with matching Placebo in period 1 (morning and evening), with Tiotropium 2.5 mcg in period 2 (morning and evening) and with a matching placebo in the morning and Tiotropium 5 mcg in the evening in period 3. All products were delivered by the Respimat inhaler, on top on maintenance therapy with iCS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Placebo/Tio R5 qd/Tio R2.5 Bid: Patients treated with a matching Placebo in period 1 (morning and evening), with a matching placebo in the morning and Tiotropium 5 mcg in the evening in period 2 and with Tiotropium 2.5 mcg in period 3 (morning and evening) . All products were delivered by the Respimat inhaler, on top on maintenance therapy with iCS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
Period: Period 1 (4 Weeks)
Arm/Group | Tio R2.5 Twice Daily (Bid) /Tio R5 Once Daily (qd) /Placebo | Tio R2.5 Bid/Placebo/Tio R5 qd | Tio R5 qd/Tio R2.5 Bid/Placebo | Tio R5 qd/Placebo/Tio R2.5 Bid | Placebo/Tio R2.5 Bid/Tio R5 qd | Placebo/Tio R5 qd/Tio R2.5 Bid
Started | 15 | 16 | 17 | 15 | 18 | 13
Completed | 15 | 15 | 16 | 15 | 16 | 12
Not Completed | 0 | 1 | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Period: Period 2 (4 Weeks)
Arm/Group | Tio R2.5 Twice Daily (Bid) /Tio R5 Once Daily (qd) /Placebo | Tio R2.5 Bid/Placebo/Tio R5 qd | Tio R5 qd/Tio R2.5 Bid/Placebo | Tio R5 qd/Placebo/Tio R2.5 Bid | Placebo/Tio R2.5 Bid/Tio R5 qd | Placebo/Tio R5 qd/Tio R2.5 Bid
Started | 15 | 15 | 16 | 15 | 16 | 12
Completed | 15 | 15 | 16 | 15 | 16 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (4 Weeks)
Arm/Group | Tio R2.5 Twice Daily (Bid) /Tio R5 Once Daily (qd) /Placebo | Tio R2.5 Bid/Placebo/Tio R5 qd | Tio R5 qd/Tio R2.5 Bid/Placebo | Tio R5 qd/Placebo/Tio R2.5 Bid | Placebo/Tio R2.5 Bid/Tio R5 qd | Placebo/Tio R5 qd/Tio R2.5 Bid
Started | 15 | 15 | 16 | 15 | 16 | 12
Completed | 15 | 15 | 16 | 15 | 16 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Total: Total number of patients randomised and treated in the study.
Arm/Group | Baseline Total
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve 0-24 Hours (AUC0-24h) Response
Description: Mixed Model Repeated Measure (MMRM) results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measurements performed in relation to evening dosing. AUC0-24h calculated using the trapezoidal rule divided by the observation time (24 hours) to report in litres.
Time Frame: 10 minutes (min) prior to first dose (baseline) and -10 min, 30 min, 60 min, 2 hours (h) , 3 h, 4 h , 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose at week 4
Population: Full Analysis Set (FAS) defined as all treated patients who had baseline data and at least 1 on-treatment efficacy measurement after 4 weeks on treatment within a period.
Measure: Mean (Standard Error); unit: L
Groups:
- Placebo: Matching Placebo bid morning and evening delivered by the Respimat inhaler, on top on maintenance therapy with iCS.
- Tio R2.5 Bid: Tiotropium 2.5 mcg bid morning and evening delivered by the Respimat inhaler, on top on maintenance therapy with iCS.
- Tio R5 qd: Tiotropium 5 mcg qd in the evening and matching placebo qd in the morning delivered by the Respimat inhaler, on top on maintenance therapy with iCS.
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.091 (0.043) | 0.241 (0.044) | 0.250 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.149, 95% CI [0.102 to 0.196], Standard Error of Mean 0.024 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.158, 95% CI [0.111 to 0.205], Standard Error of Mean 0.024 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.009, 95% CI [-0.038 to 0.056], Standard Error of Mean 0.024 — Tio R5 qd - Tio R2.5 bid

2. Secondary Outcome: Mean Pre-dose Morning Peak Expiratory Flow (PEF a.m.) Response During the Last Week on Treatment
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured by patients at home using the AM2+ device.
Time Frame: Baseline and during week 4 of each treatment period
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 88
L/min | 1.953 (5.864) | 23.281 (5.907) | 24.310 (5.924)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 21.328, 95% CI [11.084 to 31.573], Standard Error of Mean 5.190 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 22.357, 95% CI [12.044 to 32.670], Standard Error of Mean 5.225 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 1.029, 95% CI [-9.318 to 11.376], Standard Error of Mean 5.242 — Tio R5 qd - Tio R2.5 bid

3. Secondary Outcome: Mean Pre-dose Evening Peak Expiratory Flow (PEF p.m.) Response During the Last Week on Treatment
Description: as for outcome 2
Time Frame: Baseline and during week 4 of each treatment period
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 89
L/min | -1.560 (5.891) | 28.360 (5.932) | 27.096 (5.931)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 29.920, 95% CI [20.001 to 39.839], Standard Error of Mean 5.026 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 28.657, 95% CI [18.707 to 38.606], Standard Error of Mean 5.042 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -1.264, 95% CI [-11.243 to 8.716], Standard Error of Mean 5.056 — Tio R5 qd - Tio R2.5 bid

4. Secondary Outcome: FEV1 Area Under the Curve 0-12 Hours (AUC0-12h) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC0-12h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: 10 min prior to first dose (baseline) and -10 min, 30 min, 60 min, 2 h, 3 h, 4 h and 11 h 50 min related to evening dose at week 4
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.048 (0.044) | 0.217 (0.044) | 0.233 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.169, 95% CI [0.120 to 0.218], Standard Error of Mean 0.025 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.185, 95% CI [0.136 to 0.234], Standard Error of Mean 0.025 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.016, 95% CI [-0.033 to 0.065], Standard Error of Mean 0.025 — Tio R5 qd - Tio R2.5 bid

5. Secondary Outcome: FEV1 Area Under the Curve 12-24 Hours (AUC12-24h) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC12-24h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: 10 min prior to first dose (baseline) and 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose at week 4
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.135 (0.044) | 0.264 (0.045) | 0.266 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.129, 95% CI [0.077 to 0.181], Standard Error of Mean 0.026 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.131, 95% CI [0.079 to 0.183], Standard Error of Mean 0.026 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.002, 95% CI [-0.050 to 0.054], Standard Error of Mean 0.026 — Tio R5 qd - Tio R2.5 bid

6. Secondary Outcome: Peak FEV1 Within 24 Hours Post-dose Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following the evening trial-drug inhalation at the end of each 4 week period of randomised treatment.
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.337 (0.045) | 0.469 (0.045) | 0.468 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.132, 95% CI [0.084 to 0.179], Standard Error of Mean 0.024 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.131, 95% CI [0.084 to 0.179], Standard Error of Mean 0.024 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.000, 95% CI [-0.048 to 0.047], Standard Error of Mean 0.024 — Tio R5 qd - Tio R2.5 bid

7. Secondary Outcome: Trough FEV1 Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Trough FEV1 is defined as FEV1 value (performed at 10 minutes prior to the evening trial-drug inhalation) at the end of each 4 week period of randomised treatment.
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.143 (0.044) | 0.254 (0.044) | 0.275 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.111, 95% CI [0.053 to 0.170], Standard Error of Mean 0.030 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.133, 95% CI [0.074 to 0.191], Standard Error of Mean 0.029 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.021, 95% CI [-0.037 to 0.080], Standard Error of Mean 0.030 — Tio R5 qd - Tio R2.5 bid

8. Secondary Outcome: Trough Forced Vital Capacity (FVC) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Trough FVC is defined as FVC value (performed at 10 minutes prior to the evening trial-drug inhalation) at the end of each 4 week period of randomised treatment.
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.112 (0.046) | 0.179 (0.046) | 0.168 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.0515, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.068, 95% CI [0.000 to 0.136], Standard Error of Mean 0.035 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.1058, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.056, 95% CI [-0.012 to 0.124], Standard Error of Mean 0.035 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.012, 95% CI [-0.080 to 0.057], Standard Error of Mean 0.035 — Tio R5 qd - Tio R2.5 bid

9. Secondary Outcome: FVC Area Under the Curve 0-12 Hours (AUC0-12h) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following each dosing determined at the end of each 4 week treatment period. AUC0-12h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | -0.026 (0.046) | 0.099 (0.046) | 0.074 (0.046)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.125, 95% CI [0.073 to 0.177], Standard Error of Mean 0.026 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.100, 95% CI [0.048 to 0.152], Standard Error of Mean 0.026 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.025, 95% CI [-0.077 to 0.027], Standard Error of Mean 0.026 — Tio R5 qd - Tio R2.5 bid

10. Secondary Outcome: FVC Area Under the Curve 12-24 Hours (AUC12-24h) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following each dosing determined at the end of each 4 week treatment period. AUC12-24h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.032 (0.045) | 0.108 (0.045) | 0.100 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.076, 95% CI [0.023 to 0.129], Standard Error of Mean 0.027 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0123, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.068, 95% CI [0.015 to 0.120], Standard Error of Mean 0.027 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.008, 95% CI [-0.061 to 0.045], Standard Error of Mean 0.027 — Tio R5 qd - Tio R2.5 bid

11. Secondary Outcome: Peak FVC Within 24 Hours Post-dose Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following each dosing determined at the end of each 4 week treatment period.
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.302 (0.045) | 0.380 (0.045) | 0.350 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.0042, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.077, 95% CI [0.025 to 0.130], Standard Error of Mean 0.027 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0747, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.048, 95% CI [-0.005 to 0.100], Standard Error of Mean 0.027 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.029, 95% CI [-0.082 to 0.023], Standard Error of Mean 0.027 — Tio R5 qd - Tio R2.5 bid

12. Secondary Outcome: Individual FEV1 Over Time (at Each Timepoint at Visits) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L
  Timepoint -0:10 (hours:minutes) | 0.143 (0.044) | 0.254 (0.044) | 0.275 (0.044)
  Timepoint 0:30 (hours:minutes) | 0.132 (0.044) | 0.281 (0.044) | 0.304 (0.044)
  Timepoint 1:00 (hours:minutes) | 0.123 (0.044) | 0.274 (0.044) | 0.289 (0.044)
  Timepoint 2:00 (hours:minutes) | 0.103 (0.044) | 0.270 (0.044) | 0.297 (0.044)
  Timepoint 3:00 (hours:minutes) | 0.082 (0.044) | 0.264 (0.044) | 0.268 (0.044)
  Timepoint 4:00 (hours:minutes) | 0.062 (0.045) | 0.248 (0.045) | 0.263 (0.045)
  Timepoint 11:50 (hours:minutes) | -0.021 (0.049) | 0.134 (0.049) | 0.150 (0.049)
  Timepoint 12:30 (hours:minutes) | 0.075 (0.047) | 0.198 (0.047) | 0.217 (0.047)
  Timepoint 13:00 (hours:minutes) | 0.101 (0.047) | 0.250 (0.047) | 0.237 (0.047)
  Timepoint 14:00 (hours:minutes) | 0.138 (0.045) | 0.288 (0.045) | 0.282 (0.045)
  Timepoint 15:00 (hours:minutes) | 0.163 (0.046) | 0.299 (0.046) | 0.308 (0.046)
  Timepoint 16:00 (hours:minutes) | 0.161 (0.046) | 0.306 (0.046) | 0.313 (0.046)
  Timepoint 18:00 (hours:minutes) | 0.177 (0.047) | 0.300 (0.047) | 0.308 (0.047)
  Timepoint 20:00 (hours:minutes) | 0.127 (0.045) | 0.256 (0.046) | 0.245 (0.045)
  Timepoint 22:00 (hours:minutes) | 0.117 (0.047) | 0.221 (0.047) | 0.244 (0.047)
  Timepoint 23:00 (hours:minutes) | 0.124 (0.045) | 0.243 (0.045) | 0.223 (0.045)
  Timepoint 23:50 (hours:minutes) | 0.125 (0.047) | 0.232 (0.047) | 0.224 (0.047)

13. Secondary Outcome: Individual FVC Over Time (at Each Timepoint at Visits) Response
Description: as for outcome 12
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L
  Timepoint -0:10 (hours:minutes) | 0.112 (0.046) | 0.179 (0.046) | 0.168 (0.046)
  Timepoint 0:30 (hours:minutes) | 0.053 (0.047) | 0.158 (0.048) | 0.130 (0.047)
  Timepoint 1:00 (hours:minutes) | 0.055 (0.047) | 0.152 (0.047) | 0.124 (0.047)
  Timepoint 2:00 (hours:minutes) | 0.033 (0.047) | 0.131 (0.047) | 0.093 (0.047)
  Timepoint 3:00 (hours:minutes) | -0.003 (0.047) | 0.100 (0.047) | 0.057 (0.047)
  Timepoint 4:00 (hours:minutes) | -0.040 (0.049) | 0.096 (0.049) | 0.065 (0.049)
  Timepoint 11:50 (hours:minutes) | -0.064 (0.049) | 0.070 (0.049) | 0.060 (0.049)
  Timepoint 12:30 (hours:minutes) | 0.004 (0.046) | 0.133 (0.046) | 0.103 (0.046)
  Timepoint 13:00 (hours:minutes) | 0.010 (0.047) | 0.114 (0.047) | 0.102 (0.047)
  Timepoint 14:00 (hours:minutes) | 0.038 (0.047) | 0.106 (0.047) | 0.120 (0.047)
  Timepoint 15:00 (hours:minutes) | 0.034 (0.047) | 0.109 (0.047) | 0.124 (0.047)
  Timepoint 16:00 (hours:minutes) | 0.050 (0.047) | 0.111 (0.047) | 0.116 (0.047)
  Timepoint 18:00 (hours:minutes) | 0.062 (0.046) | 0.123 (0.046) | 0.113 (0.046)
  Timepoint 20:00 (hours:minutes) | 0.036 (0.047) | 0.125 (0.047) | 0.088 (0.047)
  Timepoint 22:00 (hours:minutes) | 0.028 (0.048) | 0.077 (0.048) | 0.096 (0.048)
  Timepoint 23:00 (hours:minutes) | 0.018 (0.048) | 0.094 (0.048) | 0.062 (0.048)
  Timepoint 23:50 (hours:minutes) | -0.015 (0.049) | 0.078 (0.049) | 0.052 (0.049)

14. Secondary Outcome: Individual Peak Expiratory Flow (PEF) Over Time (at Each Timepoint at Visits) Response
Description: as for outcome 12
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L/min
  Timepoint -0:10 (hours:minutes) | 19.770 (7.357) | 42.428 (7.378) | 57.897 (7.359)
  Timepoint 0:30 (hours:minutes) | 12.994 (7.275) | 46.272 (7.295) | 58.436 (7.277)
  Timepoint 1:00 (hours:minutes) | 13.783 (7.027) | 43.049 (7.043) | 53.138 (7.028)
  Timepoint 2:00 (hours:minutes) | 11.366 (7.246) | 48.328 (7.263) | 55.826 (7.248)
  Timepoint 3:00 (hours:minutes) | 9.769 (7.457) | 48.723 (7.474) | 50.747 (7.458)
  Timepoint 4:00 (hours:minutes) | 7.499 (7.242) | 42.599 (7.260) | 50.077 (7.244)
  Timepoint 11:50 (hours:minutes) | -11.219 (7.747) | 20.011 (7.765) | 26.201 (7.749)
  Timepoint 12:30 (hours:minutes) | 4.345 (7.314) | 27.436 (7.335) | 33.887 (7.316)
  Timepoint 13:00 (hours:minutes) | 6.820 (7.479) | 33.810 (7.499) | 34.582 (7.481)
  Timepoint 14:00 (hours:minutes) | 13.879 (7.323) | 44.786 (7.348) | 43.371 (7.325)
  Timepoint 15:00 (hours:minutes) | 16.125 (6.992) | 47.991 (7.012) | 45.699 (6.994)
  Timepoint 16:00 (hours:minutes) | 19.616 (7.304) | 47.697 (7.330) | 46.441 (7.306)
  Timepoint 18:00 (hours:minutes) | 20.084 (7.303) | 47.795 (7.326) | 48.790 (7.306)
  Timepoint 20:00 (hours:minutes) | 13.348 (7.213) | 42.240 (7.232) | 40.888 (7.215)
  Timepoint 22:00 (hours:minutes) | 14.275 (7.317) | 33.567 (7.339) | 41.635 (7.319)
  Timepoint 23:00 (hours:minutes) | 13.590 (7.360) | 36.712 (7.384) | 38.384 (7.362)
  Timepoint 23:50 (hours:minutes) | 15.169 (7.670) | 36.837 (7.697) | 37.595 (7.673)

15. Secondary Outcome: FVC Area Under the Curve 0-24 Hours (AUC0-24h) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. AUC0-24h calculated using the trapezoidal rule divided by the observation time (24 hours) to report in litres.
Time Frame: 10 min prior to first dose (baseline) and -10 min, 30 min, 60 min, 2 h, 3 h, 4 h , 11 h 50 min, 12 h 30 min, 13 h, 14 h, 15 h, 16 h, 18 h, 20 h, 22 h, 23 h, and 23 h 50 min related to evening dose at week 4
Population: FAS
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L | 0.003 (0.044) | 0.104 (0.044) | 0.087 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.101, 95% CI [0.055 to 0.147], Standard Error of Mean 0.023 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.084, 95% CI [0.038 to 0.130], Standard Error of Mean 0.023 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.016, 95% CI [-0.063 to 0.030], Standard Error of Mean 0.023 — Tio R5 qd - Tio R2.5 bid

16. Secondary Outcome: PEF Area Under the Curve 0-24 Hours (AUC0-24h) Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. AUC0-24h calculated using the trapezoidal rule divided by the observation time (24 hours) to report in litres/min.
Time Frame: as for outcome 15
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 90 | 89 | 90
L/min | 8.589 (6.870) | 38.831 (6.883) | 42.899 (6.871)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 30.242, 95% CI [22.167 to 38.317], Standard Error of Mean 4.091 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 34.310, 95% CI [26.240 to 42.380], Standard Error of Mean 4.089 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 4.068, 95% CI [-4.012 to 12.148], Standard Error of Mean 4.094 — Tio R5 qd - Tio R2.5 bid

17. Secondary Outcome: PEF Variability Response (Last Week on Treatment)
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. PEF variability is the absolute difference between morning and evening PEF value divided by the mean of these two values, expressed as a percent (weekly means obtained during the last week of each period of randomised treatment will be compared).
Time Frame: Baseline and during week 4
Population: FAS
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 88
Percent | 0.296 (0.711) | 0.619 (0.718) | 0.685 (0.721)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.6747, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.323, 95% CI [-1.195 to 1.841], Standard Error of Mean 0.769 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.6159, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.389, 95% CI [-1.138 to 1.916], Standard Error of Mean 0.774 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.065, 95% CI [-1.468 to 1.599], Standard Error of Mean 0.777 — Tio R5 qd - Tio R2.5 bid

18. Secondary Outcome: Mean Number of Puffs of Rescue Medication During the Whole Day (Last Week on Treatment, Response Values)
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Weekly means obtained during the last week of each period of randomised treatment will be compared.
Time Frame: Baseline and during week 4
Population: FAS
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 89
Puffs | -0.841 (0.189) | -0.917 (0.190) | -1.016 (0.190)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.5906, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.077, 95% CI [-0.358 to 0.204], Standard Error of Mean 0.142 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.2208, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.176, 95% CI [-0.458 to 0.106], Standard Error of Mean 0.143 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.099, 95% CI [-0.382 to 0.184], Standard Error of Mean 0.143 — Tio R5 qd - Tio R2.5 bid

19. Secondary Outcome: Mean Number of Puffs of Rescue Medication During Daytime (Last Week on Treatment, Response Values)
Description: as for outcome 18
Time Frame: Baseline and during week 4
Population: FAS
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 89
Puffs | -0.562 (0.106) | -0.564 (0.106) | -0.624 (0.106)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.9797, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.002, 95% CI [-0.163 to 0.159], Standard Error of Mean 0.082 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.4518, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.062, 95% CI [-0.223 to 0.100], Standard Error of Mean 0.082 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.060, 95% CI [-0.222 to 0.102], Standard Error of Mean 0.082 — Tio R5 qd - Tio R2.5 bid

20. Secondary Outcome: Mean Number of Puffs of Rescue Medication During Nighttime (Last Week on Treatment, Response Values)
Description: as for outcome 18
Time Frame: Baseline and during week 4
Population: FAS
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 88
Puffs | -0.358 (0.092) | -0.419 (0.093) | -0.432 (0.093)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.4089, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.061, 95% CI [-0.207 to 0.085], Standard Error of Mean 0.074 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.3185, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.074, 95% CI [-0.221 to 0.072], Standard Error of Mean 0.074 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.013, 95% CI [-0.160 to 0.134], Standard Error of Mean 0.074 — Tio R5 qd - Tio R2.5 bid

21. Secondary Outcome: Mean Number of Night Awakenings During the Last Week on Treatment (Score, Response Values)
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Assessed by the patient's electronic diary (eDiary incorporated in the AM2+ device), obtained during the last week of each period of randomised treatment.
Time Frame: Baseline and during week 4
Population: FAS
Measure: Mean (Standard Error); unit: Night awakenings
Arm/Group | Placebo | Tio R2.5 Bid | Tio R5 qd
Number analyzed (Participants) | 91 | 89 | 88
Night awakenings | -0.106 (0.028) | -0.104 (0.029) | -0.102 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5 Bid; Test type: Superiority or Other; p = 0.9626, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.001, 95% CI [-0.059 to 0.062], Standard Error of Mean 0.031 — Tio R2.5 bid - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.9102, Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.003, 95% CI [-0.058 to 0.065], Standard Error of Mean 0.031 — Tio R5 qd - Placebo
Statistical Analysis 3: Comparison: Tio R2.5 Bid vs Tio R5 qd; Test type: Superiority or Other; Mixed Models Analysis; MMRM adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.002, 95% CI [-0.059 to 0.063], Standard Error of Mean 0.031 — Tio R5 qd - Tio R2.5 bid

ADVERSE EVENTS:
Time Frame: 4 weeks + 30 days if in last period
Groups:
- Tio R2.5: Tiotropium 2.5 mcg bid morning and evening delivered by the Respimat inhaler, on top on maintenance therapy with iCS.
Arm/Group | Placebo | Tio R2.5 | Tio R5 qd
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/90 | 2/90
Other Adverse Events (participants affected / at risk) | 4/92 | 7/90 | 5/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | Tio R2.5 (N=90) | Tio R5 qd (N=90)
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=92) | Tio R2.5 (N=90) | Tio R5 qd (N=90)
Headache (Nervous system disorders) | 4 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.